CLINICAL TRIAL: NCT04840758
Title: A Prospective Single-arm Single-center Clinical Study：Assessment of the Safety and Effects of Stereotactic Ablation Radiotherapy (SABR) Combined With Sintilimab in Early Inoperable Synchronous Multiple Primary Lung Cancer (sMPLC)
Brief Title: Stereotactic Ablation Radiotherapy Combined With Sintilimab in Early Inoperable Synchronous Multiple Primary Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMYY-2020Y091
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Multiple Primary Lung Cancer
Keywords: Synchronous multiple primary lung cancer; inoperable; Stereotactic ablation radiotherapy; Sintilimab
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SABR+Sintilimab (Experimental): Stereotactic ablation radiotherapy (SABR) was performed sequentially on the primary and secondary lesions. Sintilimab was used 2 weeks after the end of SABR. Sintilimab : 200 mg intravenously, Q3W every cycle , given on the D1 of each cycle, and total of 4 cycles.
  Interventions: Radiation: Stereotactic Ablation Radiotherapy; Drug: Sintilimab

INTERVENTIONS:
Radiation: Stereotactic Ablation Radiotherapy — Stereotactic ablation radiotherapy was performed sequentially on the primary and secondary lesions. 50Gy/4F or 70Gy/10F were used according to the specific location of the tumor。
Drug: Sintilimab — Sintilimab was started 2 weeks after the end of radiotherapy. Sintilimab : 200 mg intravenously, Q3W every cycle , given on the D1 of each cycle, and total of 4 cycles

SUMMARY:
The purpose of this study is to assess of the Safety and Effects of Stereotactic Ablation Radiotherapy (SABR) combined with Sintilimab in early inoperable synchronous Multiple Primary Lung Cancer (sMPLC)

DETAILED DESCRIPTION:
Stereotactic ablation radiotherapy (SABR) was performed sequentially on the primary and secondary lesions. 50Gy/4F or 70Gy/10F were used according to the specific location of the tumor. Immunotherapy was started 2 weeks after the end of radiotherapy. Sintilimab : 200 mg intravenously, Q3W every cycle , given on the D1 of each cycle, and total of 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1.The diagnostic criteria for early sMPLC refer to the American College of Chest Physicians (ACCP) standard, and the following conditions should be met：

1. CT showed the presence of at least three or more lesions（Pure glass or partially solid/solid）
2. Proved to be different pathologic types by pathology.

c. If there is only one pathologically confirmed lesion or two pathological types are identical, the following conditions need to be met:

1. . The lesions are located in different lobes
2. . No mediastinal lymph node metastasis
3. . distance metastasis free

2. At least two lesions were suitable for SABR treatment.

3. ECOG performance status 0-2.

4. Stable lab values: Hematological: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets ≥100×109/L, Hemoglobin ≥9 g/dL Renal: Creatinine OR Measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤1.5× the upper limit of normal (ULN) OR ≥60 mL/min for patient with creatinine levels >1.5× institutional ULN Hepatic: Total bilirubin ≤1.5×ULN OR Direct bilirubin ≤ULN for patients with total bilirubin levels >1.5×ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN OR ≤5×ULN for patients with liver metastases ,globulin≥20 g/L, albumin≥30 g/L.

5. Female subjects must have a negative urine or serum pregnancy test within 72 hours prior to taking study drug if of childbearing potential.

6. Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

1. Previously received any T cell costimulation or immunological checkpoint treatment, including but not limited to CTLA-4 inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors or other T cell-targeting drugs.
2. An active autoimmune disease requiring systemic treatment (such as the use of disease-alleviating drugs, corticosteroids or immunosuppressants) occurred within 2 years prior to the first administration.Alternative therapies (such as thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic.
3. Interstitial lung disease, drug-induced pneumonia, radiation pneumonitis requiring steroid therapy or active pneumonia with clinical symptoms or severe pulmonary dysfunction.
4. Previous or current history of cancer other than NSCLC, except for non-melanoma skin cancer, in-situ cervical cancer or other cancers that have received curable treatment and have shown no signs of recurrence for at least 5 years.
5. Have a tendency to hereditary bleeding or coagulopathy. Clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood++ and above.
6. There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) heart failure of NYHA class 2 or higher (2) unstable angina (3) myocardial infarction within 24 weeks (4) clinical need for treatment or Interventional supraventricular or ventricular arrhythmia.
7. Uncontrolled hypertension after treatment (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90mmHg), with a history of hypertensive crisis or hypertensive encephalopathy;Uncontrolled hyperglycemia after treatment (fasting glucose >8.9mmol/L).
8. Have a history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency disease, or history of organ transplantation and bone marrow transplantation.
9. Active hepatitis B (positive detection of hepatitis B virus surface antigen [HBsAg] in the screening period, and detection of HBV-DNA detection value higher than the upper limit of the normal value of the laboratory in the research center) or hepatitis C (in the screening period, hepatitis C virus surface antibody [ HCsAb] positive, HCV-RNA positive).
10. Subjects who have received or will receive live vaccine within 30 days of the first treatment.
11. Allergic reactions to test drugs for this application.
12. The investigator determined that the subject had other factors that might lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
abscopal effect rate | at the time point of 3 Months after completion of the combined treatment
  A reaction produced following irradiation but occurring outside the zone of actual radiation absorption

SECONDARY OUTCOMES:
Incidence of Adverse events | up to approximately 1 year
  AE，according to NCI-CTCAE V4.03 and immune-related (ir) RECIST
Progression-Free Survival (PFS) | up to approximately 1 year
  PFS, defined as the time from treatment to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | up to approximately 1 year
  Disease Control Rate（DCR） according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Jiang jie, MD, Principal Investigator — First affiliated Hospital of Xiamen University

IPD SHARING:
Plan to Share IPD: No